CLINICAL TRIAL: NCT01810510
Title: Impact of PAV Versus NAVA on Patient-Ventilator Synchrony and Respiratory Muscle Unloading
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not subjects enrolled
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert Scott Harris, M.D., Associate in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013P000028
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Respiratory Failure
Keywords: respiration, artificial
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAV Ventilation (Experimental): PAV is a mode of ventilation in which the only set parameter is the proportion of work/effort that is provided regardless of the ventilatory pattern the patient chooses- the patient has full control over pressure, volume, flow and time of inspiration as well as respiratory rate. In this mode, the ventilator measures patient respiratory mechanics every 10-15 breaths and delivers a level of pressure proportional to patient effort, thereby maintaining a set proportion of patient effort regardless of the patient's ventilatory pattern. The patients will be on this mode of ventilation for 60 minutes.
  Interventions: Procedure: PAV Ventilation
- NAVA Ventilation (Experimental): With NAVA, delivery from the ventilator is triggered, controlled and cycled by the diaphragmatic EMG signal (Edi), which is measured by a specially designed nasogastric or orogastric catheter (NGT or OGT) containing EMG electrodes that cross the diaphragm. In this mode, the ventilator measures the Edi with each breath and instantaneously delivers a level of pressure proportional to Edi magnitude, thereby providing a set proportion of effort on a breath-to-breath basis. The patients will be on this mode of ventilation for 60 minutes.
  Interventions: Procedure: NAVA Ventilation

INTERVENTIONS:
Procedure: PAV Ventilation — PAV is a mode of ventilation in which the only set parameter is the proportion of work/effort that is provided regardless of the ventilatory pattern the patient chooses- the patient has full control over pressure, volume, flow and time of inspiration as well as respiratory rate. In this mode, the ventilator measures patient respiratory mechanics every 10-15 breaths and delivers a level of pressure proportional to patient effort, thereby maintaining a set proportion of patient effort regardless of the patient's ventilatory pattern. The patients will be on this mode of ventilation for 60 minutes.
  Arms: PAV Ventilation
Procedure: NAVA Ventilation — With NAVA, delivery from the ventilator is triggered, controlled and cycled by the diaphragmatic EMG signal (Edi), which is measured by a specially designed nasogastric or orogastric catheter (NGT or OGT) containing EMG electrodes that cross the diaphragm. In this mode, the ventilator measures the Edi with each breath and instantaneously delivers a level of pressure proportional to Edi magnitude, thereby providing a set proportion of effort on a breath-to-breath basis. The patients will be on this mode of ventilation for 60 minutes.
  Arms: NAVA Ventilation

SUMMARY:
The purpose of this study is to determine whether two modes of artificial (i.e. mechanical) ventilation have an impact on patient synchrony with the ventilator (breathing machine) and on the patient's work of breathing.

DETAILED DESCRIPTION:
New, "intelligent" ventilator modes with more complex closed loops have been developed, some with a demonstrated clinical benefit. The modes of proportional assist ventilation (PAV) and neurally-adjusted ventilatory assist (NAVA) are capable of delivering ventilation proportional to patient effort and may be associated with improved patient-ventilator synchrony when compared to pressure support ventilation (PSV), a classic simple closed-loop assisted ventilation mode.

This study will study both modes of ventilation (PAV and NAVA) in each patient who is recruited, and measures of patient-ventilator synchrony and work of breathing will be taken during each mode.

Baseline data will be collected on a standardized volume-cycled control mode ventilator setting for 5 minutes and on a standardized pressure support ventilator mode for 25 minutes. Subjects will then be randomized to either PAV or NAVA ventilation and will be ventilated on that mode for 30 minutes. Equivalence of support levels between PAV and NAVA trials will be ensured by targeting the same peak (Ppeak) airway pressures. Data collected will include (but are not limited to) vital signs, sedation score, dyspnea assessment using visual analog scale, respiratory rate, tidal volume (Vt), peak airway pressure (Ppeak), inspiratory time and neural inspiratory time (Ti and Tni), total physiologic and neural respiratory cycle time (Ttot and Tntot), end-tidal CO2, esophageal pressure waveforms, waveforms of all ventilatory patterns, Edi waveforms, and peak Edi. Subjects will then be switched to the other mode of ventilation and undergo an identical 30-minute evaluation period with identical data collection. Arterial blood gas measurements will be done after any changes in ventilator settings only in subjects who have had arterial lines inserted for clinically-indicated reasons. This will be a replicate crossover study, meaning that all subjects that are initially randomized to one sequence (PAV-NAVA or NAVA-PAV) will afterwards be "crossed-over" to the other one. These two additional periods of measurements will allow us to account for potential carry over effects of the different interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Respiratory failure requiring mechanical ventilation
* Spontaneously breathing (able to generate flow/ pressure/ volume triggers on control modes of ventilation or on a mode of mechanically assisted spontaneous breathing)
* Requiring FiO2< 60% and PEEP< 10cm H2O to maintain oxygen saturations >90%

Exclusion Criteria:

* Pregnancy
* Inability to tolerate spontaneous breathing
* Gastro-esophageal pathology (including but not limited to recent gastric or esophageal surgery, history of varices, known anatomical gastric or esophageal defects such as strictures, hernias or fistulas)
* Agitation necessitating major sedative infusions
* Hemodynamic instability necessitating active adjustments in vasopressor therapy
* Coagulopathy
* New intracranial pathology (stroke, hemorrhage, meningitis, encephalitis)
* Paralyzed diaphragm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patient-Ventilator Synchrony | 2.5 hours
  Patient-ventilator synchrony will be assessed during both modes of ventilation. Data collected will include (but is not limited to) vital signs, sedation score, respiratory rate, tidal volume (Vt), peak airway pressure (Ppeak), inspiratory time and neural inspiratory time (Ti and Tni), total physiological and neural respiratory cycle time (Ttot and Tntot), waveforms of all ventilatory patterns, end-tidal CO2, esophageal pressure waveforms, Edi waveforms, and peak Edi.

SECONDARY OUTCOMES:
Dyspnea Index | 2.5 hours
  Patients who are able to interact (i.e. who are sufficiently awake and attentive) will undergo a dyspnea assessment, including a visual analogue scale for dyspnea.
Respiratory Muscle Unloading | 2.5 hours
  Respiratory muscle unloading, i.e. reduction of work of breathing by the patient, will be assessed during both modes of ventilation. Data collected will include (but is not limited to) vital signs, sedation score, respiratory rate, tidal volume (Vt), peak airway pressure (Ppeak), inspiratory time and neural inspiratory time (Ti and Tni), total physiological and neural respiratory cycle time (Ttot and Tntot), waveforms of all ventilatory patterns, end-tidal CO2, esophageal pressure waveforms, Edi waveforms, and peak Edi.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Harris, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States